CLINICAL TRIAL: NCT04257513
Title: Innovative Therapeutic Strategy Targeting Neurons with Cholesterol in Huntington Disease: from Preclinical Studies to Clinical Trial Readiness
Brief Title: Clinical Study to Monitor Plasma Levels of 24OHC in Subject with HD
Acronym: Chol-HD
Status: Completed | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Other Study IDs: Chol-HD
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; Cholesterol
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy controls subjects: Subjects without known family history of HD, or tested negative for the HD expansion mutation.
  Interventions: Diagnostic Test: Brain MRI
- Symptomatic HD subjects: Subjects HD gene expansion carriers who have clinical diagnostic motor symptoms of defined HD, and disease stage I to III.
  Interventions: Diagnostic Test: Brain MRI
- Presymptomatic HD subjects:: Subjects HD gene expansion carriers who not have clinical diagnostic motor features of HD.
  Interventions: Diagnostic Test: Brain MRI

INTERVENTIONS:
Diagnostic Test: Brain MRI — Neurological and Cognitive evaluation; Brain MRI

SUMMARY:
A 2-year clinical longitudinal study to measure plasma concentrations of 24S-hydroxycholesterol, a brain-derived cholesterol catabolite, in subjects with Huntington disease, from the presymptomatic to the symptomatic stages.

DETAILED DESCRIPTION:
In cross-sectional studies, the plasma level of brain-derived 24S-hydroxycholesterol (24OHC) has been found to be significantly diminished in HD patients from the first stages of the disease. Furthermore, in HD gene-positive pre-symptomatic (pre-HD) the plasma levels can predict the development of motor signs of disease in subjects closer to onset, better than in subjects far from onset. These data suggest that circulating 24OHC might be a candidate biomarker for phenotypic conversion and for disease progression in different stages of the disease.

Detailed neurological, cognitive and imaging data and blood samples will be collected at baseline, and after two years to investigate the rate of changes along the longitudinal study. Isotope dilution mass spectrometry (assay performed at Istituto di Ricerche Farmacologiche Mario Negri IRCCS) will be used to measure the plasma levels of brain-derived 24OHC and other sterols reflecting peripheral cholesterol synthesis. The investigators expect to establish whether changes in plasma 24OHC mark disease progression and, eventually, phenoconversion from pre-symptomatic to symptomatic stages in combination with clinical, cognitive and imaging parameters.

ELIGIBILITY:
Inclusion Criteria:

Symptomatic HD subjects

1. Age ≥ 18 years
2. Known family history of HD and genetically confirmed disease by direct DNA test (CAG expansion > 35 repeats)
3. Clinical diagnostic motor features of HD, defined as score> 5 at the motor Unified Huntington Disease Rating Scale (mUHDRS)
4. Stage I or II or III HD, defined as UHDRS Total Functional Capacity (TFC) scores between 3 and 13 inclusive (Marder, 2000)

Presymptomatic HD subjects

1. Age ≥ 18 years
2. Known family history of HD and genetically confirmed mutation by direct DNA test (CAG expansion > 35 repeats)
3. Absence of clinical motor features of HD, defined as mUHDRS rating scale ≤ 5

Healthy Subjects

1. Age ≥ 18 years
2. Absence of known family history of HD or genetically confirmed negative DNA test for HD (CAG expansion ≤ 35 repeats)
3. Absence of clinical motor features of HD, defined as mUHDRS rating scale ≤ 5

Exclusion Criteria:

1. Participation in clinical pharmacological trials
2. Inability to undergo and tolerate MRI scans (e.g. claustrophobia, severe chorea, MRI-incompatible intrauterine devices, metal implants, ect)
3. Inability or unwillingness to undertake any of the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 60 subjects (both males and females) will be enrolled in the study. Eligible participants include healthy controls, people who are in the presymptomatic stage of HD, and people with symptomatic HD at different disease stage (I-III).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
plasmatic 24OHC levels | at baseline and after 2-years follow up visit
  Changes in plasmatic 24OHC levels measured

SECONDARY OUTCOMES:
Changes in the score of the Unified Huntington Disease Rating Scale (UHDRS) | after 2-years follow up visit
  The concentration of 24OHC will be correlated with clinical evaluation to the stage of the disease and its progression.
Changes in score at the Digit Symbol Modalities Test (DSMT) | after 2-years follow up visit
  The concentration of 24OHC will be correlated with cognitive evaluation to the stage of the disease and its progression.
Changes in caudate nucleus volume measured at MRI | after 2-years follow up visit
  The concentration of 24OHC will be correlated with Imaging the stage of the disease and its progression.

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Genetica Medica e Neurogenetica, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No